CLINICAL TRIAL: NCT01837160
Title: The Identification of In Vivo Angiogenesis and Fibrosis in Aortic Stenosis Using Positron Emission Tomography
Brief Title: Angiogenesis and Fibrosis in Aortic Stenosis
Status: Completed | Type: Observational
Sponsor: University of Edinburgh (Other)
Responsible Party: Sponsor
Other Study IDs: 2012/R/CAR/23; FS/12/84/29814 (Other Grant/Funding Number: BHF Clinical Research Training Fellowship)
Record Dates: First submitted 2013-03-14; First posted 2013-04-23 (Estimated); Last update posted 2016-08-30 (Estimated); Status verified 2015-03

CONDITIONS: Aortic Stenosis; Fibrosis; Neovascularization, Pathologic
Keywords: Angiogenesis; Fibrosis; Aortic Stenosis; Imaging; CT-PET; PET-CT; Cardiac MRI
MeSH Terms: conditions — Aortic Valve Stenosis; Fibrosis; Neovascularization, Pathologic | interventions — Transcatheter Aortic Valve Replacement

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood samples will be taken, and the serum frozen and stored for further analysis pending ethical approval.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (5):
- Healthy Volunteers: 10 patients with normal echocardiogram studies and no history of ischaemic heart disease.
  Patients to recieve CT-PET with fluciclatide, cardiac MRI scan, CT-coronary angiogram and echocardiogram.
  Interventions: Procedure: Cardiac MRI scan; Radiation: CT-PET scan; Procedure: Echocardiogram; Radiation: CT-coronary angiogram scan
- Moderate Aortic Stenosis (n=10): Patients with moderate aortic stenosis. Patients are to recieve Cardiac MRI, CT-PET scan, echocardiography and CT-coronary angiogram scan at baseline.
  They will undergo repeat cardiac MRI scan and echocardiogram at 12 - 24 months.
  Interventions: Procedure: Cardiac MRI scan; Radiation: CT-PET scan; Procedure: Echocardiogram; Radiation: CT-coronary angiogram scan
- Mild Aortic Stenosis (n=10): Patients with mild aortic stenosis. Patients are to recieve Cardiac MRI, CT-PET scan, echocardiography and CT-coronary angiogram scan at baseline.
  They will undergo repeat cardiac MRI scan and echocardiogram at 12 - 24 months.
  Interventions: Procedure: Cardiac MRI scan; Radiation: CT-PET scan; Procedure: Echocardiogram; Radiation: CT-coronary angiogram scan
- Severe aortic Stenosis (n=10): Patients with severe aortic stenosis. Patients are to recieve Cardiac MRI, CT-PET scan, echocardiography and CT-coronary angiogram scan at baseline.
  They will undergo repeat cardiac MRI scan and echocardiogram at 12 - 24 months.
  Interventions: Procedure: Cardiac MRI scan; Radiation: CT-PET scan; Procedure: Echocardiogram; Radiation: CT-coronary angiogram scan
- Severe Aortic Stenosis for AVR (n=10): Patients with severe aortic stenosis proceeding to aortic valve replacement. Patients are to recieve Cardiac MRI, CT-PET scan, echocardiography and CT-coronary angiogram scan at baseline.
  They will undergo a repeat CT-PET scan 3 months after the operation.
  They will undergo repeat cardiac MRI scan and echocardiogram at 12 months after the operation.
  Interventions: Procedure: Cardiac MRI scan; Radiation: CT-PET scan; Procedure: Echocardiogram; Radiation: CT-coronary angiogram scan; Procedure: Aortic Valve Replacement

INTERVENTIONS:
Procedure: Cardiac MRI scan — Cardiac MRI scan with assessment of late gadolinium enhancement and T1 mapping.
Radiation: CT-PET scan — Computed Tomography / Positron Emission Tomography scan with 18F-fluciclatide tracer.
Procedure: Echocardiogram — Echocardiography.
Radiation: CT-coronary angiogram scan — CT-coronary angiogram following CT-PET scan. Standard protocol.
Procedure: Aortic Valve Replacement — For AVR (already scheduled prior to enrollment)
  Other Names: AVR
  Groups: Severe Aortic Stenosis for AVR (n=10)

SUMMARY:
Angiogenesis and fibrosis lie at the heart of a number of fundamental processes responsible for cardiovascular disease. In this proposal, the investigators intend to build upon a highly successful programme of studies exploring the cardiovascular applications of positron emission tomography. Specifically, the investigators will explore the potential role of a novel radiotracer, 18F-fluciclatide, which is a highly selective ligand for the αvβ3 and αvβ5 integrin receptors that are up regulated during angiogenesis, and tissue fibrosis and remodelling. This tracer has been successfully used to assess angiogenesis in metastatic tumours and its uptake is suppressed by anti-angiogenic therapies. The investigators here propose to describe the pattern of uptake of 18F-fluciclatide in cardiovascular diseases, specifically aortic stenosis and aortic atherosclerosis. The investigators will correlate 18F-fluciclatide uptake with in vivo measures of angiogenesis and fibrosis as well as ex vivo histological characterisation of tissue. If successful, this novel radiotracer could provide an extremely important non-invasive method of assessing in vivo angiogenesis, plaque vulnerability, and tissue remodelling as well as potential applications in developing stem cell therapies.

DETAILED DESCRIPTION:
Integrins

Integrins are a group of molecules responsible for intercellular adhesion and signalling. They comprise a superfamily of heterodimeric receptors that are composed of 18 different α and β subunits. In combination, they can generate 24 different receptor subtypes with a range of physiological and pathophysiological functions. The αvβ3 receptor is an integrin that is found at low levels on mature endothelial cells but is markedly up regulated on endothelial cells of actively growing blood vessels. It was previously known as the vitronectin receptor although it was subsequently found to bind many other ligands including fibrinogen, fibronectin, laminin, thrombospondin, von Willebrand factor, and certain collagen subtypes. These features are also seen with the αvβ5 integrin receptor, with both receptors recognising the arginine-glycine-aspartate (RGD) motif present on these ligands.

1.1.2 Role of αvβ3 and αvβ5 Integrins in Cardiovascular Disease

The expression of αvβ3 and αvβ5 receptors is up regulated in a number of diseased states and this has been particularly well characterised in the angiogenesis associated with tumour growth and metastases. However, there are many potential roles for this integrin pathway in cardiovascular disease including myocardial infarction, atherosclerosis, restenosis, aortic stenosis and aneurysm disease that have been relatively unexplored.

1.1.2.1 Aortic Stenosis

Aortic stenosis is characterized by extensive valvular thickening due to accumulation of fibrous tissue and remodeling of the extracellular matrix. In all three layers of the valve, abundant fibroblast-like cells are found and are commonly referred to as valvular interstitial cells. A sub-population of these cells become activated by the inflammatory activity within the valve and differentiate into myofibroblasts. Whilst fibroblasts control the synthesis of collagen in the normal valve, myofibroblasts are responsible for the accelerated fibrosis observed within stenotic valves. In addition, matrix metalloproteinases are secreted by myofibroblasts and inflammatory cells, and have an important and complex role in the restructuring of the valve leaflet matrix. As already indicated, activation and differentiation of fibroblasts into myofibroblasts are dependent on αvβ3 and αvβ5 receptor expression. In addition, mirroring the situation in carotid atherosclerosis, patients with severe aortic stenosis have a high incidence (78%) of intraleaflet haemorrhage and this is associated with angiogenesis and more rapid disease progression.

Histopathological studies have confirmed fibrosis to be an integral part of the left ventricular hypertrophic process in aortic stenosis. Myofibroblasts infiltrate the myocardium and secrete extracellular matrix proteins including collagen types I and III. Areas of fibrosis are observed to co-localize with areas of myocyte apoptosis and it has been suggested that fibrosis occurs as a form of scarring after myocyte death and injury. As with fibrosis in the valve, the renin-angiotensin system, transforming growth factor-beta and an imbalance in matrix metalloproteinase and their tissue inhibitor activity have all been implicated in this process. A mid-wall pattern of fibrosis has been observed in the myocardium of up to 38% of patients with moderate or severe aortic stenosis and has been associated with a more advanced hypertrophic response. Importantly, there is also an 8-fold increase in mortality associated with mid-wall fibrosis.

1.1.2.2 Atherosclerosis and Restenosis

The development of atherosclerosis is due to a complex interplay of oxidised lipid, inflammatory cell infiltration, and smooth muscle cell migration in the arterial wall. Once established, atherosclerotic plaques may progress and rupture leading to the clinical presentations of acute myocardial infarction and stroke. Features associated with plaque rupture include a thin fibrous cap, lipid-rich pool and intraplaque haemorrhage. Indeed, plaque rupture is particularly associated with plaque neovascularisation and vascular-endothelial growth factor expression suggesting that instability may be induced by angiogenesis. Thus, up regulation of αvβ3 and αvβ5 receptors may represent a novel marker of, and potential therapeutic target for, plaque vulnerability.

1.1.3 Fluciclatide

Fluciclatide is a RGD-containing cyclic peptide that has recently been developed as an 18F-radiotracer to detect tumour angiogenesis by positron emission tomography. It is highly selective for the αvβ3 and αvβ5 receptors with affinities (EC50) of 11.1 and 0.1 nM respectively with minimal cross reactivity with the αIIbβ3 receptor (EC50 281 nM). Pre-clinical tumour work has demonstrated that 18F-fluciclatide is taken up by glioblastomas and that this is suppressed by the anti-angiogenic tyrosine kinase inhibitor, sunitinib, confirming the specificity of fluciclatide for areas of angiogenesis. It has been assessed in phase I clinical trials and found to be safe and well tolerated.

1.1.4 Aims

To date, there have been many preclinical studies examining the application of radiotracers targeting the αvβ3 and αvβ5 integrin receptors. The clinical application of these tracers has been largely limited to oncology as a method of assessing angiogenesis within tumours. Here we wish to explore the role of the αvβ3 and αvβ5 receptor radiotracer, 18F-fluciclatide, to assess angiogenesis and fibrosis in patients with aortic stenosis as a measure of both valvular and myocardial fibrosis. This patient group will have co-existent aortic atheroma and this will provide us with an opportunistic assessment of tracer uptake in atherosclerosis. We feel it is important to assess a range of cardiovascular conditions to determine whether αvβ3 and αvβ5 integrin receptor expression is particular to certain disease processes. If successful, these preliminary data will permit the more detailed exploration of specific disease areas and novel therapeutic interventions. At present, fluciclatide is not licensed or approved for clinical use and is being used here as an Investigational Agent to explore the pathophysiology of aortic stenosis.

1.2 ORIGINAL HYPOTHESES

We hypothesise that 18F-fluciclatide can identify the expression of the αvβ3 and αvβ5 integrin receptors in vivo in man in two major cardiovascular disease areas: aortic atherosclerosis and aortic stenosis. Specifically, we hypothesise that 18F-fluciclatide will:

1. Be taken up into aortic atherosclerotic plaque.
2. Show demonstrable uptake in the aortic valve and myocardium of patients with aortic stenosis that will correlate with the degree of active angiogenesis and fibrosis.

6.1 ANGIOGENESIS AND FIBROSIS IN AORTIC STENOSIS

Aortic stenosis is associated with substantial left ventricular hypertrophy and consequent myocardial fibrosis with the latter predicting prognosis. Left ventricular hypertrophy and associated fibrosis is also a major risk factor for adverse cardiovascular events in a number of other conditions including essential hypertension. Cardiac magnetic resonance imaging is the gold-standard method of assessing for the presence of myocardial fibrosis but it does not necessarily indicate the on going activity of the fibrotic process. In this study, we will assess the uptake of 18F-fluciclatide in patients with aortic stenosis as a model of pressure overload left ventricular hypertrophy. We will also seize the opportunity to determine whether there is any uptake of 18F-fluciclatide in the aortic valve given that this has been shown to have areas of fibrosis and angiogenesis.

All study patients and healthy volunteers will undergo blood sampling, echocardiogram, positron emission and computed tomography scans with 18F-fluciclatide as well as cardiac magnetic resonance imaging with assessment of gadolinium late enhancement. Following injection of 18F-fluciclatide, patients will be monitored using our standard clinical approach, including observation of haemodynamic parameters, and this will continue throughout their study visit until departure. In patients undergoing aortic valve replacement surgery, aortic valve tissue will be retained and a 3-mm tru-cut biopsy of left ventricular myocardium obtained with which to compare the findings from the scans.

Healthy volunteer patients will not undergo repeat assessment. After a period of one to two years from their initial scan, patients with Aortic Stenosis will return for repeat blood sampling, cardiac magnetic resonance imaging with assessment of late gadolinium enhancement and echocardiogram. Those patients who have undergone an aortic valve replacement will undergo repeat positron emission and computed tomography scans with 18F-fluciclatide six months after their operation, prior to their second cardiac MRI scan.

Blood samples will be assessed using standard clinical biochemical and haematological profiles such as full blood count and urea and electrolytes. In addition, markers of cardiac ischaemia, fibrosis and angiogenesis will be assessed. Additional serum, plasma and DNA will be stored at -80 degrees Celsius for future potential analyses.

6.1.2 Study Interpretation

We anticipate that myocardial uptake of 18F-fluciclatide will be increased in patients with aortic stenosis and left ventricular hypertrophy. We expect the degree of myocardial uptake to correlate with cardiac magnetic resonance imaging assessment of fibrosis as well as the histological measures of fibrosis and αvβ3 and αvβ5 integrin receptor expression. We expect the degree of myocardial uptake to predict cardiac magnetic resonance imaging assessment of fibrosis following a period of one to two years. In exploratory analyses, we will also take the opportunity to assess the extent of 18F-fluciclatide uptake within the aortic valve itself, and if successful, correlate this with histological measures of angiogenesis and fibrosis.

6.2 ANGIOGENESIS IN AORTIC ATHEROSCLEROSIS

Patients with aortic stenosis will have a high prevalence of concomitant aortic atherosclerosis. In Dr Dweck's Fellowship, we were able to exploit this association and undertake secondary analyses of 18F-sodium fluoride uptake in aortic and coronary atherosclerosis. This generated some highly innovative findings that informed our understanding of atherosclerosis and the role of calcification.

6.2.1 Study Schedule

We will use the datasets obtained from the patients above to explore the uptake of 18F-fluciclatide within the thoracic aorta. Atherosclerosis will be identified using computed tomography and magnetic resonance images obtained of the thorax at the time of the study scans. No additional image acquisition will be required. This will provide pilot data to inform subsequent dedicated studies focused on acutely inflamed atherosclerotic plaques, such as patients with recent transient ischaemic attacks or strokes attributable to carotid disease.

ELIGIBILITY:
Inclusion Criteria

* asymptomatic mild (peak valve velocity of 2-5-3.0 m/s; n=10), moderate (peak valve velocity of 3.0-4.0 m/s; n=10) or severe aortic stenosis (peak valve velocity of >4.0 m/s; n=10) and 10 patients with severe aortic stenosis proceeding to aortic valve replacement.
* Healthy control subjects (n=10) will have no past medical history of ischaemic heart disease or valvular heart disease and have a structurally normal heart on echocardiography.

Exclusion Criteria:

* Atrial fibrillation
* Hepatic failure (Childs-Pugh grade B or C)
* Renal failure (estimated glomerular filtration rate <25 mL/min)
* Women of child-bearing potential
* Contraindication to magnetic resonance imaging
* Inability to undergo scanning
* Ochronosis and those with any form of collagen-vascular disease.

Min Age: 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 50 patients in total, recruited from Cardiology Outpatient Clinics
Sampling Method: Non-Probability Sample
Enrollment: 21 (Actual)
Dates: Start 2013-04; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
The mean and maximum standardised uptake values (SUV) of fluciclatide for the myocardium and its correlation with the severity of aortic stenosis determined echocardiographically. | 1 - 2 years
The mean and maximum standardised uptake values (SUV) of fluciclatide for the myocardium and its correlation with the volume of myocardial fibrosis on magnetic resonance scanning. | 1 - 2 years

SECONDARY OUTCOMES:
The mean and maximum standardised uptake values (SUV) of fluciclatide in the aortic valve in patients with aortic stenosis | 1 year
The mean and maximum standardised uptake values (SUV) of fluciclatide in concomitant aortic atheroma | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: David E Newby, MBChB PhD, Study Director — University of Edinburgh; William Sa Jenkins, MBChB MRCP, Principal Investigator — University of Edinburgh
Locations (1):
- University of Edinburgh, Edinburgh, Lothian, United Kingdom